CLINICAL TRIAL: NCT01404208
Title: 2/2 D-Cycloserine Augmentation of CBT for Pediatric OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of South Florida (Other)
Responsible Party: Principal Investigator, Daniel A. Geller, M.D., Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011P000875; 1R01MH093402-01A1 (NIH)
Record Dates: First submitted 2011-07-25; First posted 2011-07-27 (Estimated); Results first posted 2017-02-27 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-02

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D-Cycloserine (Active Comparator)
  Interventions: Drug: D-Cycloserine
- Sugar Pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D-Cycloserine — 25mg dose for children weighing between 22.5kg and 45kg (dose = approx. .7mg/kg) 50mg dose for children weighing greater than 46kg (dose = approx. .7mg/kg) Dose given 7 times, every seven days, except for the third dose, which will be given three days after the second dose. All doses given 1 hour prior to therapy session.
  Arms: D-Cycloserine
Drug: Placebo — Sugar pill
  Arms: Sugar Pill

SUMMARY:
The purpose of this study is to find out if D-Cycloserine (DCS), taken at the same time as a child gets cognitive behavioral therapy (CBT) can help children with pediatric obsessive-compulsive disorder.

Cognitive Behavior Therapy is a talking therapy that will teach children new skills to better cope with his/her OCD. CBT usually uses "exposure-based therapy". This means that the person with OCD slowly learns to deal with things they usually avoid. This is done by moving from less stressful situations to more challenging ones.

The investigators hope to enroll about 75 children ages 7-17 years old with OCD in this study at Massachusetts General Hospital (MGH). The National Institute of Mental Health (NIMH) is paying for this study to be done.

If your child qualifies for the study, the investigators will assign him or her by chance (like a coin toss) to either the DCS group or the placebo group. You and the study doctor cannot choose your child's study group. Your child will have an equal chance (1 in 2) of being assigned to the DCS group.

Your child will be asked to take one or two capsules of the study drug (either DCS or placebo, depending which study group they were assigned to) one hour before CBT visits 4-10. The study coordinator will give your child the study drug at the location of the CBT sessions. This is to make sure that your child takes the study drug one hour before his/her scheduled therapy session. We will ask you to record any bad side effect from the study drug that your child may have before each CBT session.

It will take your child about 34 weeks to complete the study. During this time, the investigators will ask you and your child to make a minimum of 17 trips to the study center. There may be up to 23 trips when including CBT Booster sessions.

This study uses a placebo. The placebo looks exactly like the DCS, but it contains no DCS. The investigators use placebos in research studies to learn if the the results are caused by the study drug or are due to other reasons. This is a double-blind study. A double-blind study is a study where both the doctor and the study participant do not know whether the study participant is being given DCS or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Obsessive-Compulsive Disorder as primary or co-primary diagnosis
* Score on CY-BOCS of 16 or greater
* Full Scale IQ greater than or equal to 85
* English speaking

Exclusion Criteria:

* Receiving concurrent psychotherapy or a past adequate trial of CBT for OCD
* Initiation of an antidepressant within 12 weeks before study enrollment
* Initiation of an antipsychotic within 6 weeks before study enrollment
* No new alternative medications, nutritionals, or therapeutic diets within 6 weeks of study enrollment
* Any change in established psychotropic medication within 8 weeks before study enrollment (6 weeks for antipsychotic). Alternative medications must be stable for 6 weeks prior to baseline. Any medications must remain stable during treatment.
* Current clinically significant suicidality
* Suicidal behaviors within six months
* DSM-IV conduct disorder
* DSM-IV autism
* DSM-IV bipolar
* DSM-IV schizophrenia or schizo-affective disorders
* Substance abuse within the past six months
* Hoarding symptoms (due to difficulty implementing E/RP tasks)
* Weight less than 22.5k
* Epilepsy or renal insufficiency
* Current and/or past history of alcohol abuse (DCS is contraindicated)
* Pregnant or having unprotected sex (in females)
* Presence of a significant and/or unstable medical illness that might lead to hospitalization during the study
* Known DCS allergy

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 206 (Actual)
Dates: Start 2011-07; Primary Completion 2015-09 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Geller, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Storch EA, Murphy TK, Goodman WK, Geffken GR, Lewin AB, Henin A, Micco JA, Sprich S, Wilhelm S, Bengtson M, Geller DA. A preliminary study of D-cycloserine augmentation of cognitive-behavioral therapy in pediatric obsessive-compulsive disorder. Biol Psychiatry. 2010 Dec 1;68(11):1073-6. doi: 10.1016/j.biopsych.2010.07.015. PMID 20817153
- See also: The OCD and Related Disorder Program at Massachusetts General Hospital — https://mghocd.org/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 206 subjects were initially enrolled at MGH and USF. Of those, 32 were considered screen fails and 32 were not randomized either because they did not meet inclusion or exclusion criteria at randomization or because they withdrew consent or dropped out. Thus, 142 participants were randomized.
Period: Overall Study
Arm/Group | D-Cycloserine | Sugar Pill
Started | 70 | 72
Completed | 67 | 72
Not Completed | 3 | 0
Not completed — Discontinued | 3 | 0

BASELINE CHARACTERISTICS:
Population: 206 subjects were initially enrolled at MGH and USF. Of those, 32 were considered screen fails and 32 were not randomized either because they did not meet inclusion or exclusion criteria at randomization or because they withdrew consent or dropped out. Thus, 142 participants were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | D-Cycloserine | Sugar Pill | Total
Number analyzed (Participants) | 70 | 72 | 142
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.67 (2.94) | 12.14 (2.97) | 12.40 (2.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 34 | 76
  Male | 28 | 38 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 10 | 22
  Not Hispanic or Latino | 58 | 62 | 120
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 61 | 65 | 126
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS)
Description: The CY-BOCS is a measure of severity of OCD symptoms, including interference, time spent on thoughts or behaviors, distress, resistance, etc. The CY-BOCS is measured from 0 to 40, with larger values indicating more severe symptoms. Our outcome measure was the difference between the post treatment and randomization scores. When those values are negative, it indicates a reduction in symptom severity.
Time Frame: Change from Score at Randomization to Post Treatment
Measure: Mean (Standard Deviation); unit: Change in score from randomization
Arm/Group | D-Cycloserine | Sugar Pill
Number analyzed (Participants) | 70 | 72
Change in score from randomization | -10.35 (7.72) | -9.40 (7.05)

2. Secondary Outcome: Clinical Global Impression-Severity (CGI-Severity)
Description: The Clinical Global Impression-Severity is a 7-point clinician rating of illness severity, with a score of 0 indicating no illness and a score of 6 indicating extremely severe symptoms. Because the secondary outcome was the change in score from randomization to post treatment, a more negative score indicates a greater reduction in symptom severity.
Time Frame: Change from Randomization Point to Post Treatment
Measure: Mean (Standard Deviation); unit: Change in score from randomization
Arm/Group | D-Cycloserine | Sugar Pill
Number analyzed (Participants) | 70 | 72
Change in score from randomization | -1.39 (1.04) | -1.2 (.91)

ADVERSE EVENTS:
Arm/Group | D-Cycloserine | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/72
Other Adverse Events (participants affected / at risk) | 60/70 | 70/72
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | D-Cycloserine (N=70) | Sugar Pill (N=72)
Headache (Nervous system disorders) | 39 | 33
Constipation (Gastrointestinal disorders) | 17 | 9
Poor Memory (Nervous system disorders) | 19 | 8
Nausea or Vomiting (Gastrointestinal disorders) | 23 | 25
Feeling Drowsy or Sleepy (General disorders) | 27 | 28
Blurred Vision or Reading (Eye disorders) | 8 | 7
Increased Appetite (Metabolism and nutrition disorders) | 17 | 13
Difficulty Starting Urination (Renal and urinary disorders) | 7 | 5
Trouble Concentrating (Nervous system disorders) | 23 | 26
Nightmares (Nervous system disorders) | 16 | 11
Difficulty Sitting Still (General disorders) | 19 | 23
Heartbeat Irregular or Pounding (Cardiac disorders) | 9 | 7
Diarrhea (Gastrointestinal disorders) | 16 | 11
Frequent Need to Urinate (Renal and urinary disorders) | 14 | 4
Dry Mouth (General disorders) | 17 | 13
Decreased Appetite (Metabolism and nutrition disorders) | 17 | 9
Tremors or Shakiness (General disorders) | 11 | 8
Skin Rash or Irritation (Skin and subcutaneous tissue disorders) | 11 | 13
Ringing in the Ears (Ear and labyrinth disorders) | 9 | 7
Sweating (Skin and subcutaneous tissue disorders) | 12 | 15
Faintness or Lightheadedness (Nervous system disorders) | 18 | 13
Poor Coordination (General disorders) | 11 | 9
Stiffness in the Muscles (Musculoskeletal and connective tissue disorders) | 14 | 10
Trouble Falling Asleep (General disorders) | 31 | 28
Feeling Tired (General disorders) | 32 | 29
Waking up During the Night (General disorders) | 24 | 17
Waking up too Early in the Morning (General disorders) | 18 | 17
Feeling Confused (Nervous system disorders) | 14 | 8
Feeling Nervous or Sad (Psychiatric disorders) | 27 | 21
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 20 | 13
Ear infection (Ear and labyrinth disorders) | 2 | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 | 7
Coughing (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Stomach pain or discomfort (Gastrointestinal disorders) | 4 | 9
Mouth or dental pain (General disorders) | 0 | 4
Fever (General disorders) | 1 | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Body abrasions and bruising (Injury, poisoning and procedural complications) | 4 | 1
Anxiety (Psychiatric disorders) | 7 | 2
Seasonal Allergies (Immune system disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No